CLINICAL TRIAL: NCT06686381
Title: A Phase II, Randomized, Non-comparative Double Arm, Open-label, 2-stage, Multicenter Study to Evaluate the Efficacy and Safety of 2 Tetra-modality Bladder Preservation Strategies in Muscle-invasive Bladder Cancer With Maximum TURBT Followed by Induction Platinum-based Chemotherapy/Avelumab Followed by Radiation Therapy Then Maintenance Avelumab or Watch and Wait Approach
Brief Title: Tetra-modality Bladder Preservation Strategies in Muscle-invasive Bladder Cancer: TURBT+ Chemo/Immunotherapy+ Radiation Therapy+ Maintenance Immunotherapy vs. W&W
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2024-0290
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Muscle-invasive Bladder Cancer
Keywords: Muscle-invasive bladder cancer; Bladder preservation; Avelumab; Tetramodalities
MeSH Terms: interventions — Drug Therapy; Radiotherapy; Watchful Waiting; Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a non-comparative, randomized trial, where each arm is independent from the other. Arm A will receive drug A in both the induction and maintenance phases, while Arm B will receive drug A during the induction phase and then follow a "watch and wait" approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Maintenance Avelumab) (Experimental): Arm A: TURBT followed by induction Chemo/immunotherapy (DDMVAC (6 cycles) + Avelumab (6 cycles) or cisplatin/Gemzar (4 cycles) + Avelumab (6 cycles). A clinical evaluation is scheduled at 4 months post-day1 cycle 1 with CT scan/MRI for chest/abdomen/pelvis (CTCAP), Cystoscopy with Biopsy and urine cytology. Then complete or near complete responders will undergo 20 fractions of hypo-fractionated radiotherapy 55 grays followed by Avelumab every 2 weeks for 12-month maintenance phase.
  Interventions: Procedure: Maximum TURBT; Drug: Chemotherapy + Immunotherapy Induction; Radiation: Radiotherapy; Drug: Immunotherapy Maintenance
- Arm B (W&W) (Experimental): Arm B: TURBT followed by induction Chemo/immunotherapy (DDMVAC (6 cycles) + Avelumab (6 cycles) or cisplatin/Gemzar (4 cycles) + Avelumab (6 cycles). A clinical evaluation is scheduled at 4 months post-day1 cycle 1 with CT scan/MRI for chest/abdomen/pelvis (CTCAP), Cystoscopy with Biopsy and urine cytology. Then complete or near complete responders will undergo 20 fractions of hypo-fractionated radiotherapy 55 grays followed by 1 year watch and wait.
  Interventions: Procedure: Maximum TURBT; Drug: Chemotherapy + Immunotherapy Induction; Radiation: Radiotherapy; Other: Watchful waiting with supportive care

INTERVENTIONS:
Procedure: Maximum TURBT — Total removal of the bladder tumor through TURBT
Drug: Chemotherapy + Immunotherapy Induction — Chemotherapy: DDMVAC (6 cycles) or Gemcitabine-Cisplatin (4 cycles) Immunotherapy: Avelumab (6 cycles)
Radiation: Radiotherapy — Hypofractionated radiotherapy: 20 fractions, 55 Grays
Drug: Immunotherapy Maintenance — Maintenance Avelumab every 2 weeks for 12 months
  Arms: Arm A (Maintenance Avelumab)
Other: Watchful waiting with supportive care — 1 year watch and wait
  Arms: Arm B (W&W)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of adding the immunotherapy Avelumab as a fourth component, alongside tumor removal, chemotherapy, and radiation, to increase the chance of preserving the bladder in the treatment of muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
Muscle-invasive bladder cancer (MIBC) is an aggressive form of bladder cancer, with a 5-year survival rate of about 40%.

The standard treatment for MIBC is induction platinum-based chemotherapy followed by radical cystectomy. Recently bladder preservation strategies have emerged as an alternative to radical cystectomy, particularly useful for patients who are unfit for surgery or would rather opt for non-surgical approaches. Knowing the high risks related to surgery and its significant complications, the investigators propose to implement 2 tetra-modalities treatment strategies to increase the chance of preserving the bladder and decrease the need of salvage cystectomy.

The purpose of this study is to assess the efficacy and safety of 2 bladder-preservation treatments plans called tetra-modalities:

First plan:

* maximium TURBT
* chemo-immunotherapy as induction phase (Avelumab added to chemotherapy)
* radiation therapy
* maintenance phase with Avelumab

Second plan:

* Maximum TURBT
* chemo-immunotherapy as induction phase (Avelumab added to chemotherapy)
* radiation therapy
* Watch and wait

Both tetra-modalities duration will last maximum of 2 years from patient inclusion.

These treatment plans are based on the synergistic action between immunotherapy, chemotherapy, and radiotherapy. The use of Avelumab in the maintenance group is supported by its proven success in treating advanced cancer and various studies looking at immunotherapy as a way to avoid or delay bladder removal.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF) before any trial related procedures.
2. Male or female participant with ≥ 18 years of age at time of consenting.
3. Participant is able and willing to comply with the requirements of trial protocol.
4. Pathologically (histologically or cytologically) and radiologically confirmed newly diagnosed MIBC (T2-T4 N0 M0) or recurrent previously NMIBC.
5. Histologically confirmed transitional cell carcinoma.
6. Participant with ECOG Performance Status (PS) ≤ 1 at screening visit.
7. An estimated life expectancy of more than 6 months.
8. At screening visit, Left Ventricular Ejection Fraction LVEF >50% by echocardiography, for participants planned to receive DDMVAC.
9. Participant must have adequate laboratory values at screening visit as follow:

   1. Hematologic:

      * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
      * Platelet count ≥ 100 × 10^9/L
      * Hemoglobin ≥ 9 g/dL (may have been transfused)
   2. Hepatic:

      * Total bilirubin level ≤ 1.5 × ULN
      * AST ≤ 2.5 × ULN
      * ALT ≤ 2.5 × ULN
   3. Renal:

      * Estimated creatinine clearance > 50 mL/min according to the Cockcroft-Gault formula
      * Serum urea ≤ 1.5 x ULN
      * Serum creatinine ≤ 1.5 x ULN.
10. Female participant of childbearing potential must have a negative serum pregnancy test at screening.
11. For female participant of childbearing potential: use one of the following highly effective contraception methods throughout the trial and for 30 days after the last Avelumab treatment administration.

    * combined (estrogen and progesterone) hormonal contraception associated with inhibition of ovulation: either oral, intravaginal or transdermal
    * progesterone-only hormonal contraception associated with inhibition of ovulation: either oral, injectable or implantable
    * intrauterine device (IUD)
    * intrauterine hormone-releasing system (IUS)
    * bilateral tubal occlusion
    * vasectomised partner (provided that partner is the sole sexual partner of the female trial participant and that the vasectomised partner has received medical assessment of the surgical success)
    * sexual abstinence

Exclusion Criteria:

1. Participant with non-muscle invasive bladder cancer or Metastatic disease (M1) and/or lymph node positive.
2. Participant who underwent radical cystectomy or is planned for radical cystectomy.
3. Histologically confirmed squamous cell carcinoma, micropapillary carcinoma, neuroendocrine carcinoma, adenocarcinoma, or mixed histology.
4. Participant had received treatment for urothelial carcinoma, with any of the following anti-cancer therapies prior the first dose of trial treatment: systemic chemotherapy, targeted small molecule therapy, or radiation therapy.
5. Participant had received prior treatment with any drug or antibody (anti-PD-1, anti-PD- L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody) targeting T-cell co-stimulation or checkpoint pathways.
6. Participant who are not eligible to receive DDMVAC or Cisplatin-Gemzar.
7. History of severe hypersensitivity to Avelumab or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI- CTCAE v5.0 Grade ≥ 3).
8. Participant with hydronephrosis.
9. Active infection requiring systemic therapy within 28 days before the first dose of trial treatment (e.g., urinary tract infection).
10. History of testing positive for the human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
11. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening visit (positive Hepatitis B surface antigen (HBsAg) or HCV RNA if anti-HCV antibody screening test is positive).
12. Participant currently using immunosuppressive medication, except for the following:

    * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection).
    * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent.
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
13. Active autoimmune diseases that might deteriorate upon receiving an immune- stimulatory agent. Conditions such as vitiligo, psoriasis, diabetes type I, or hypo - or hyper-thyroid diseases not requiring immunosuppressive treatment are eligible.
14. Participant has any of the following medical conditions: Addison's disease, thyroiditis/Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, and Grave's disease.
15. Any psychiatric condition that would prohibit the understanding or rendering of informed consent form.
16. Hepatic insufficiency manifesting as clinical jaundice, hepatic encephalopathy, and/or variceal bleed within 60 days prior to screening.
17. Clinically significant, active cardiovascular disease, such as:

    * Transmural myocardial infarction within 6 months of enrollment
    * Unstable angina
    * Congestive heart failure (New York Heart Association Classification Grade II or greater)
    * Serious cardiac arrhythmia requiring medical treatment
18. Cerebral vascular accident/ stroke within 6 months of enrollment.
19. End-stage renal disease requiring dialysis.
20. Participant has severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior.
21. Prior organ transplantation including allogenic stem-cell transplantation.
22. Treatment with an investigational agent within 28 days before the first dose of trial treatment.
23. Participation in another clinical trial.
24. Participants who are taking prohibited medication.
25. Pregnant or breastfeeding women or who are planned to get pregnant or breastfeed during the trial.
26. Vaccination within 4 weeks of the first dose of Avelumab is prohibited except for administration of inactivated vaccines.
27. Persisting toxicity related to prior therapy with Grade > 1 (NCI-CTCAE v 5.0); with the exception of: alopecia, sensory neuropathy Grade ≤ 2, or other toxicity with Grade ≤ 2 not constituting a safety risk based on investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Avelumab in 2 non-comparative arms | 2 years
  2 years proportion of MIBC bladder preserved participants in each tetra-modality arm.

SECONDARY OUTCOMES:
Response rate post-induction | At week 17 (after 4 months of induction)
  Response rate of participants in each arm following induction chemo/immunotherapy
Quality of life | Every 3 weeks (up to 3 months), then every 4 months (up to 1 year)
  Effect of each tetra-modality arm on the quality of life of participants using the Functional Assessment of Cancer Therapy - Bladder (FACT-Bl) questionnaire; FACT-Bl total score range: 0-156 (higher scores mean worse quality of life)
Safety | During treatment (up to 90 days after end of treatment)
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shamseddine A, Abbas N, Temraz S, Al Darazi M, Charafeddine M, Dagher K, Youssef B, Nasr R, Khauli R, El Hajj A, Bulbul M. Tetra-modality bladder preservation with avelumab for muscle-invasive urothelial cancer: a phase II trial (TRIUMPH-B01). Future Oncol. 2025 Dec;21(30):3873-3884. doi: 10.1080/14796694.2025.2549244. Epub 2025 Aug 25. PMID 40851456